CLINICAL TRIAL: NCT06178484
Title: Comparison of Surgical Repair Versus Functional Treatment in Patients With Proximal ACL Tear
Acronym: SUTUFONC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS-2022-12-063
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: ACL - Anterior Cruciate Ligament Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Functional treatment: Functional treatment combines the use of splints, rehabilitation and muscle strengthening
- Surgical treatment: Surgical treatment means ACL tear repair

SUMMARY:
Isolated ruptures of the anterior cruciate ligament (ACL) can be proximal, distal or occur in the middle of the ACL.

Treatment of patients with proximal lesions should be graded. Functional treatment can be reserved for low-demanding patients in whom the practice level is limited and the risk of progression to a knee functionally unstable less marked. In athletes, the risk of a new sprain must be explained and the patient will choose a functional treatment or a surgical treatment.

Few studies exist in the literature on the superiority of surgical treatment compared to functional treatment. In this context, this study is based on the hypothesis that patients undergoing ACL surgical repair have better functional scores and more intense sport activity than patients with functional treatment.

DETAILED DESCRIPTION:
Isolated ruptures of the anterior cruciate ligament (ACL) are ligament injuries which lead to the most surgical interventions on the capsuloligamentous system of the knee. These ruptures can be proximal, distal or occur in the middle of the ACL.

Treatment of patients with proximal lesions should be graded and should take into account patient's symptoms (feeling of instability), physical examination data, amount of residual ligament, sport practice, practice level, time interval since the initial trauma, work requirements… Functional treatment can be reserved for low-demanding patients in whom the practice level is limited and the risk of progression to a knee functionally unstable (positive pivot shift) less marked. In athletes, the risk of a new sprain must be explained and the patient will choose a functional treatment or a surgical treatment.

Functional treatment is variable, combining the use of splints, rehabilitation, muscle strengthening. The healing time is three months. Wearing a splint has not proven its effectiveness in preventing progression to rupture complete when resuming sporting activities. If instability is revealed, it is then necessary move towards ACL reconstruction treatment.

Surgical treatment generally involves ligamentoplasty at the expense of a knee tendon to replace the ruptured ACL. In the context of ACL proximal tear, the patient may be offered surgical repair of the ACL.

There are many studies on the results of ACL ligamentoplasties but literature is poor on the outcomes of modern ACL repairs. Surgical repair of the proximal rupture of ACL has experienced renewed interest in recent years thanks to the appearance of new fixing systems. Used in the 70s and 80s, this technique was gradually little abandoned in the mid-1980s following disappointing results in favor autograft reconstruction techniques.

Few studies exist in the literature on the superiority of surgical treatment compared to functional treatment. In this context, this study is based on the hypothesis that patients undergoing ACL surgical repair have better functional scores and more intense sport activity than patients with functional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient with no history of knee surgery except meniscal surgery
* Patient whose period is less than 3 months between the date of the accident and the surgery
* Patient with an isolated proximal Sherman 1 or 2 ACL tear
* Patient with a proximal Sherman 1 or 2 ACL tear associated to a stable meniscal lesion or to an MCL or LCL lesion grade 1 or 2 but not grade 3
* Patient practicing a non-contact pivot sport (sliding sports, board sports,racket)

Exclusion Criteria:

* Patient with contralateral ACL tear
* Patient practicing a pivot sport with contacts
* Patient presenting external rotary jumps ++ and +++
* Patient with an ACL tear Sherman 3 or 4
* Patient with meniscal lesions in the shape of a bucket handle or tabs unstable meniscals
* Patient with a surgical history on the knee concerned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACL tear treated with functional or surgery treatment
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective IKDC (International Knee Documentation Committee) score | 1 day
  Subjective IKDC score is based on 10 questions linded to knee status. This score is ranging from 0 to 100. 100 means a level of sport activity and daily activity without any limit in the absence of any symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé La Louvière, Lille, Choisir Une Région, France

IPD SHARING:
Plan to Share IPD: No